CLINICAL TRIAL: NCT00179439
Title: Nasal Potential Difference Testing: Evaluation of Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) Function in Children With Primary Sclerosing Cholangitis (PSC)
Brief Title: NPDT Evaluation in Children With CFTR and (PSC)
Acronym: NPD
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Steven Freedman, MD PhD Full Professor Harvard Medical School, Beth Israel Deaconess Medical Center
Other Study IDs: 2004P-000316; 02820-4
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Primary Sclerosing Cholangitis; Inflammatory Bowel Disease
Keywords: PSC; IBD; CFTR
MeSH Terms: conditions — Cholangitis, Sclerosing; Inflammatory Bowel Diseases

INTERVENTIONS:
Procedure: nasal potential difference testing

SUMMARY:
The investigators hypothesize that PSC in children is associated with mutations and functional changes of the cystic fibrosis (CF) gene.

DETAILED DESCRIPTION:
The purpose of this protocol is to perform Nasal Transepithelial Potential Difference (NTPD) testing to assess the function of the cystic fibrosis gene product, a chloride channel referred to as CFTR, in patients diagnosed with PSC and/or inflammatory bowel disease in childhood and currently 12 years of age and greater.

Dr. Freedman's laboratory has shown that there is an increased prevalence of CFTR abnormalities in adults with PSC as demonstrated by genotype and phenotype analysis. We hypothesize that abnormalities in CFTR based on exhaustive genotype and phenotype assessments are associated with the presence of PSC in children. We would like to enroll patients with inflammatory bowel disease and no PSC to use as a "control group".

Subjects with PSC and/or inflammatory bowel disease diagnosed in childhood, currently aged 12 years and above, will be enrolled in study protocols at Children's Hospital in Boston, which will have received their local IRB approval. The only role for BIDMC will be to perform NTPD testing on these subjects. No other assessment or testing will be performed at our site. We will not be involved in any other aspect of care for these subjects.

ELIGIBILITY:
Inclusion Criteria:

* 12 years of age and older
* Must have diagnosis of primary sclerosing cholangitis and/or inflammatory bowel disease
* Absence of other liver disease, such as viral hepatitis, drug-induced liver disease, and metabolic/hereditary liver disease
* No exclusion based on sex, race, and ethnic background

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-01 (Actual); Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
CFTR DNA analysis

SECONDARY OUTCOMES:
Nasal potential difference testing
Sweat test

CONTACTS AND LOCATIONS:
Overall Officials: Harpreet Pall, MD, Study Director — Boston Children's Hospital; Steven D Freedman, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States